CLINICAL TRIAL: NCT06658626
Title: An Open-label Phase 1 Study to Evaluate Metabolism, Excretion, and Mass Balance of [¹⁴C]MK-0616 in Healthy Participants
Brief Title: A Study to Evaluate the Metabolism, Excretion, and Mass Balance of [¹⁴C]Enlicitide Chloride ([¹⁴C]MK-0616) in Healthy Participants (MK-0616-016)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 0616-016; MK-0616-016 (Other: MSD)
Record Dates: First submitted 2024-10-24; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Healthy
MeSH Terms: interventions — MK-0616

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [¹⁴C]Enlicitide chloride (Experimental): Participants will receive a single dose of [¹⁴C]enlicitide chloride on Day 1.
  Interventions: Drug: [¹⁴C]Enlicitide chloride

INTERVENTIONS:
Drug: [¹⁴C]Enlicitide chloride — IV Injection
  Other Names: MK-0616

SUMMARY:
The purpose of this study is to learn what happens to enlicitide chloride labeled with [¹⁴C] in a person's body over time. A label can be added to a study medicine to trace it in a person's body.

ELIGIBILITY:
Inclusion Criteria:

* Is in good health.
* Has a body mass index ≥18 and ≤32 kg/m^2, inclusive.

Exclusion Criteria:

* Has a history of cancer.
* Has positive tests for hepatitis B surface antigen, hepatitis C antibodies or human immunodeficiency virus.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2023-03-10 (Actual); Primary Completion 2023-08-02 (Actual); Study Completion 2023-08-02 (Actual)

PRIMARY OUTCOMES:
Cumulative Amount of Radioactivity Excreted in Urine (Aeu) | At designated timepoints (up to 15 days)
  Urine samples will be collected to determine the Aeu of [¹⁴C]enlicitide chloride.
Cumulative Amount of Radioactivity Excreted in Feces (Aef) | At designated timepoints (up to 15 days)
  Fecal samples will be collected to determine the Aef of [¹⁴C]enlicitide chloride.
Cumulative Percentage of Radioactivity Excreted in Urine (feu) | At designated timepoints (up to 15 days)
  Urine samples will be collected to determine the feu of [¹⁴C]enlicitide chloride.
Cumulative Percentage of Radioactivity Excreted in Feces (fef) | At designated timepoints (up to 15 days)
  Fecal samples will be collected to determine the fef of [¹⁴C]enlicitide chloride.
Plasma Enlicitide Chloride: Area Under the Concentration-Time Curve from Time 0 to the Last Measurable Concentration (AUC0-t) | At designated timepoints (up to 15 days)
  Plasma samples will be collected to determine the AUC0-t of enlicitide chloride.
Plasma Enlicitide Chloride: Area Under the Concentration-Time Curve from Time 0 to Infinity (AUC0-inf) | At designated timepoints (up to 15 days)
  Plasma samples will be collected to determine the AUC0-inf of enlicitide chloride.
Plasma Enlicitide Chloride: Maximum Plasma Concentration (Cmax) | At designated timepoints (up to 15 days)
  Plasma samples will be collected to determine the Cmax of enlicitide chloride.
Plasma Enlicitide Chloride: Apparent Terminal Half-life (t1/2) | At designated timepoints (up to 15 days)
  Plasma samples will be collected to determine the t1/2 of enlicitide chloride.
Plasma Enlicitide Chloride: Time to Maximum Plasma Concentration (Tmax) | At designated timepoints (up to 15 days)
  Plasma samples will be collected to determine the Tmax of enlicitide chloride.
Plasma Total Reactivity: AUC0-t | At designated timepoints (up to 15 days)
  Plasma samples will be collected to determine the AUC0-t of total reactivity.
Plasma Total Reactivity: AUC0-inf | At designated timepoints (up to 15 days)
  Plasma samples will be collected to determine the AUC0-inf of total reactivity.
Plasma Total Reactivity: Cmax | At designated timepoints (up to 15 days)
  Plasma samples will be collected to determine the Cmax of total reactivity.
Plasma Total Reactivity: t1/2 | At designated timepoints (up to 15 days)
  Plasma samples will be collected to determine the t1/2 of total reactivity.
Plasma Total Reactivity: Tmax | At designated timepoints (up to 15 days)
  Plasma samples will be collected to determine the Tmax of total reactivity.
Enlicitide Chloride to Total Radioactivity Ratio of Area Under the Concentration-Time Curve from Time 0 to the Last Detectable Sample (enlicitide chloride AUC0-x/total radioactivity AUC0-x) | At designated timepoints (up to 15 days)
  Plasma samples will be collected to determine the enlicitide chloride AUC0-x/total radioactivity AUC0-x.

SECONDARY OUTCOMES:
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 29 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of the study intervention, whether or not considered related to the study intervention.
Number of Participants Who Discontinue the Study Due to an AE | Up to approximately 29 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of the study intervention, whether or not considered related to the study intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Labcorp Clinical Research Unit Inc. (Site 0001), Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com